CLINICAL TRIAL: NCT05989711
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Pemvidutide in Non-Cirrhotic Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: IMPACT TRIAL: Efficacy and Safety of Pemvidutide in Subjects With Nonalcoholic Steatohepatitis (NASH)
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT- 801-203
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pemvidutide 1.2 mg (n=38) (Experimental)
  Interventions: Drug: Pemvidutide
- Pemvidutide 1.8 mg (n=76) (Experimental)
  Interventions: Drug: Pemvidutide
- Placebo (n=76) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pemvidutide — Administered by subcutaneous injection
  Arms: Pemvidutide 1.2 mg (n=38); Pemvidutide 1.8 mg (n=76)
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo (n=76)

SUMMARY:
Purpose of this study is to assess the effects of pemvidutide on NASH resolution and NASH fibrosis.

DETAILED DESCRIPTION:
A Phase 2, multi-center, double-blind, placebo-controlled study to evaluate the efficacy and safety of pemvidutide in NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female 18-75 years
3. Histologic diagnosis of NASH and/or histologic confirmation of NASH based on central pathology evaluation of a liver biopsy during screening

   1. A histologic NAFLD Activity Score (NAS) ≥ 4 with a score of at least 1 on each subcomponent score based on central pathology evaluation (steatosis [0-3], lobular inflammation [0-3], and hepatocyte ballooning [0-2])
   2. NASH fibrosis stages 2 through 3 according to the NASH CRN fibrosis staging system based on central pathology evaluation
4. Subject agrees to have a liver biopsy performed during the screening period (if no biopsy within the preceding 6 months is available) and at 24 weeks of treatment
5. BMI ≥ 27.0 kg/m2
6. Subjects with Type 2 diabetes mellitus (T2D) should be on a stable treatment regimen for their T2D for at least 90 days prior to screening
7. Subject meets at least 3 of the 5 criteria of Metabolic Syndrome (American Heart Association 2005)
8. Liver fat content by MRI-PDFF ≥ 8%

Exclusion Criteria:

1. Weight gain or loss > 5% in the 3 months prior to randomization or > 10% in the 6 months prior to screening
2. History or clinical evidence of Type 1 diabetes mellitus
3. Hemoglobin A1c (HbA1c) > 9.5% or clinically significant persistent hyperglycemia
4. Liver conditions:

   1. History of cirrhosis or complications of cirrhosis, including but not limited to variceal bleeding, encephalopathy, or ascites
   2. Documented causes of chronic liver disease other than NASH
   3. ALT or AST laboratory values > 5 × ULN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving NASH resolution (NAFLD activity score [NAS], ballooning = 0; lobular inflammation = 0, 1) with at least a 2-point reduction in NAS without worsening of fibrosis | 24 weeks
Proportion of subjects achieving at least 1 stage improvement in liver fibrosis without worsening of NASH (defined as no change in the NAS, ie, the sum score for ballooning, inflammation, and steatosis) | 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects achieving the composite of both NASH resolution and at least 1 stage improvement of liver fibrosis at 24 weeks | 24 weeks
Relative change (%) in liver fat content by MRI-PDFF | 24 weeks and 48 weeks
Absolute change in MRI-based corrected T1 (cT1) imaging | 24 weeks and 48 weeks
Absolute change in alanine aminotransferase (ALT) | 24 weeks and 48 weeks
Absolute change in Enhanced Liver Fibrosis (ELF) score | 24 weeks and 48 weeks
Absolute change in Fibroscan-AST (FAST) score | 24 weeks and 48 weeks
Relative (%) change in body weight | 24 weeks and 48 weeks
Absolute changes in fasting lipids (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides) | 24 weeks and 48 weeks
Change in HbA1c (%) | 24 weeks and 48 weeks
Change in glucose (mg/dL) | 24 weeks and 48 weeks
Change in systolic and diastolic blood pressure (mmHg) | 24 weeks and 48 weeks
Change in heart rate (beats per minute) | 24 weeks and 48 weeks
The number of subjects with treatment emergent adverse events | 48 weeks

CONTACTS AND LOCATIONS:
Locations (38):
- United States (27):
  - Altimmune Clinical Study Site, Chandler, Arizona
  - Altimmune Clinical Study Site, Peoria, Arizona
  - Altimmune Clinical Study Site, Tucson, Arizona
  - Altimmune Clinial Study Site, Tucson, Arizona
  - Altimmune Clinical Study Site, North Hollywood, California
  - Altimmune Clinical Study Site, Panorama City, California
  - Altimmune Clinical Study Site, Englewood, Colorado
  - Altimmune Clinical Study Site, Bradenton, Florida
  - Altimmune Clinical Study Site, Fort Myers, Florida
  - Altimmune Clinical Study Site, Hialeah Gardens, Florida
  - Altimmune Clinical Study Site, Miami Lakes, Florida
  - Altimmune Clinical Study Site, Port Orange, Florida
  - Altimmune Clinical Study Site, Sarasota, Florida
  - Altimmune Clinical Study Site, West Palm Beach, Florida
  - Altimmune Clinical Study Site, Dalton, Georgia
  - Altimmune Clinical Study Site, Marietta, Georgia
  - Altimmune Clinical Study Site, Bastrop, Louisiana
  - Altimmune Clinical Study Site, Shreveport, Louisiana
  - Altimmune Clinical Study Site, Clarksville, Tennessee
  - Altimmune Clinical Study Site, Germantown, Tennessee
  - Altimmune Clinical Study Site, Austin, Texas
  - Altimmune Clinical Study Site, Bellaire, Texas
  - Altimmune Clinical Study Site, Edinburg, Texas
  - Altimmune Clinical Study Site, Georgetown, Texas
  - Altimmune Clinical Study Site, Houston, Texas
  - Altimmune Clinical Study Site, San Antonio, Texas
  - Altimmune Clinical Study Site, West Jordan, Utah
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital/ Translational Research Institute, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Box Hill Hospital, Box Hill, Victory
  - Monash Hospital, Clayton, Victory
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Altimmune Clinical Study Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Noureddin M, Harrison SA, Loomba R, Alkhouri N, Chalasani N, Sheikh MY, Tomah S, Gutierrez JA, Urbina S, Suschak JJ, Brown R, Odili O, Yang J, Keeton S, Neff G, Mena E, Roberts MS, Browne SK, Harris MS. Safety and efficacy of weekly pemvidutide versus placebo for metabolic dysfunction-associated steatohepatitis (IMPACT): 24-week results from a multicentre, randomised, double-blind, phase 2b study. Lancet. 2025 Dec 6;406(10520):2644-2655. doi: 10.1016/S0140-6736(25)02114-2. Epub 2025 Nov 11. PMID 41237796